CLINICAL TRIAL: NCT05023317
Title: Multi-site Pilot Trial of Strengths-based Linkage to Alcohol Care (SLAC) for Hazardous Drinkers in Primary Care
Brief Title: Strengths-based Linkage to Alcohol Care (SLAC) for Hazardous Drinkers in Primary Care
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 20-058
Record Dates: First submitted 2021-08-17; First posted 2021-08-26 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Alcohol-induced Disorders; Alcohol Drinking; Mental Health
Keywords: referral and consultation; psychosocial intervention
MeSH Terms: conditions — Alcohol-Induced Disorders; Alcohol Drinking; Psychological Well-Being | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two conditions-(a) strengths based linkage to alcohol care plus usual care or (b) usual care only
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research assistants, blinded to condition, will collect baseline and 3-month follow-up data from participants. The investigators will also be blinded to participant group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strengths-based linkage to alcohol care (SLAC) (Experimental): SLAC is a behavioral intervention designed to link persons with substance use/misuse to a care or help option
  Interventions: Behavioral: Strengths-based linkage to alcohol care
- Usual care (Active Comparator): Usual care consists of brief intervention in primary care and/or standard referral to more intensive alcohol care (e.g., outpatient/inpatient, pharmacotherapy)
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Strengths-based linkage to alcohol care — SLAC is a behavioral intervention designed to link persons with substance use/misuse to care
  Other Names: SLAC
  Arms: Strengths-based linkage to alcohol care (SLAC)
Behavioral: Usual care — Usual care consists of brief screening and intervention and/or standard referral to alcohol care
  Arms: Usual care

SUMMARY:
This pilot study will determine the feasibility, acceptability, and efficacy of Strengths-based Linkage to Alcohol Care (SLAC; a behavioral intervention) to link Veterans, identified as hazardous drinkers in VHA primary care, to alcohol care. Participants screening positive in VA primary care for hazardous drinking and posttraumatic stress disorders (PTSD) and/or depression in the past year will be recruited. Participants will be randomly assigned to one of two study conditions - SLAC plus usual care or usual care only. The investigators will determine the feasibility of conducting a larger scale study to evaluate SLAC in primary care and SLAC's acceptability among key stakeholders (e.g., Veterans, primary care providers). Other outcomes will include exploring whether SLAC improves linkage to an alcohol care or help option and/or reduces alcohol use and mental health (PTSD, depression) symptoms.

DETAILED DESCRIPTION:
Background: It is important for Veterans with hazardous drinking to link to evidence-based alcohol care given high rates of comorbid mental health symptoms (PTSD, depression). Veterans with symptoms of PTSD who engage in hazardous drinking are at high risk for developing more severe drinking problems and depression. And Veterans with PTSD or depression are three to four times more likely to report hazardous drinking than Veterans without either of these disorders. This project will determine the feasibility, acceptability, and efficacy of Strengths-based Linkage to Alcohol Care (SLAC) to link Veterans, identified as hazardous drinkers in VHA primary care (PC), to alcohol care.

Significance/Impact: Existing VHA options, referral by a PC provider or mental health provider co-located in PC, for linking Veterans with hazardous drinking in PC to alcohol care are largely ineffective. Therefore, this proposal directly addresses HSR&D priorities in the areas of Access to Care, Mental Health, and Primary Care by testing a novel approach to linking Veterans engaging in hazardous drinking, in the PC setting, to VA and non-VA alcohol care, to improve their drinking and mental health outcomes.

Innovation: This project is highly innovative because it offers a solution to the critical gap in VHA care in which PC patients with hazardous drinking are not receiving alcohol care. It tests a strategy to increase linkage to alcohol care that is both intensive enough to produce change, yet feasible to use in busy clinical settings with too-high demand on too-few staff members. In addition, the intervention proposed (SLAC) targets Veterans with the entire spectrum of hazardous drinking, including those with mental health symptoms. A highly innovative feature of SLAC is that it teaches PC providers how to link Veterans to evidence-based alcohol care instead of teaching providers how to treat hazardous drinking in the PC setting. Providers' lack of knowledge on how to treat hazardous alcohol use is a substantial obstacle to Veterans receiving alcohol care. Additional unique and innovative features of SLAC are that it uses patients' self-identified strengths, abilities, and skills to help them link to alcohol care.

Specific Aims: (Aim 1): To adapt SLAC for use among Veterans with hazardous drinking who may also have comorbid mental health symptoms, and for delivery by telephone in the VHA PC setting. The investigators will conduct qualitative interviews with Veterans, PC staff, and the VACO partners to ensure that the content and format of SLAC are adapted so they are relevant and acceptable to these stakeholders. (Aim 2): To determine (a) the feasibility of conducting a larger scale randomized controlled trial (RCT) to test SLAC's effectiveness and (b) SLAC's acceptability among hazardous drinking Veterans in PC, and to explore (c) the efficacy of SLAC among hazardous drinking Veterans in PC. To achieve Aim 2, the investigators will conduct a multi-site pilot RCT of SLAC at two VA medical facilities (Little Rock, AR and Palo Alto, CA). To achieve Aims 2a-b, the investigators will measure the feasibility (e.g., rates of enrollment and follow-up, fidelity to the SLAC intervention) of conducting a subsequent larger RCT (to test SLAC's effectiveness) and SLAC's acceptability (SLAC completion rates, satisfaction with SLAC) among Veterans. To achieve Aim 2c, the investigators will explore the efficacy of SLAC to improve Veterans' linkage and engagement in alcohol care, and their alcohol and mental health outcomes, at 3-month follow-up.

Methodology: The investigators will use (Aim 1) qualitative interviews to adapt SLAC for Veterans and for the PC setting, and (Aim 2) conduct a multi-site, pilot RCT.

Implementation/Next Steps: Should the findings justify a subsequent project, the investigators plan to propose a fully powered, multi-site study, using a Hybrid design, to test SLAC's clinical effectiveness when delivered in VHA PC while observing and gathering information on the implementation potential of SLAC in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Have screened positive for hazardous drinking (AUDIT-C score > 5)
* PTSD (PC-PTSD-5 score > 3) and/or depression (PHQ-2 score > 3) in the prior 12 months and have positive rescreens
* Not have received specialty SUD treatment or participated in weekly mutual-help groups in the past 90-days
* Not have significant cognitive impairment
* Have ongoing access to a mobile or landline telephone
* Provide at least one contact who will know the Veteran's contact information

Exclusion Criteria:

* Not meeting any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Linkage to alcohol care | 3-month
  This outcome is a dichotomous variable (yes/no), with "yes" defined as the participant reporting at least one of the following: attended an initial meeting with an outpatient (primary care, specialty care) or residential program; attended a mutual-help group meeting; received > 30-days' supply of AUD medication; or went online to access e-health for alcohol information.
Utilization of alcohol care | 3-month
  The investigators will define utilization as the percentage of days, in the past 90-days, that participants obtained any alcohol care.
Utilization of alcohol care options | 3-month
  We will measure the total number of alcohol care options participants obtained over the past 90-days; scores will range from 0 (no care) to 4 (obtained all types of care: outpatient/residential, mutual-help, medication (>30-days' supply), e-health).

SECONDARY OUTCOMES:
Alcohol consumption | 3-month
  The quantity and frequency of alcohol consumed will be measured using the 90-day Time Line Follow-Back (TLFB) instrument. The TLFB is a calendar that tracks alcohol consumed each day. We will combine frequency data (days of alcohol consumed) and quantity data (number of drinks consumed each day) to derive a variable measuring harmful drinking days - or days in which alcohol consumed is above NIAAA recommended limits for men and women.
Depression | 3-month
  Depression severity will be measured using the Patient Health Questionnaire-9. Scores range from 0-27. Higher scores indicate more symptoms of depression.
Posttraumatic stress disorder | 3-month
  Posttraumatic stress disorder severity will be measured using the PTSD Checklist-5. Scores range from 0-80, with higher scores indicating more symptoms of PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Cucciare, PhD, Principal Investigator — Central Arkansas Veterans Healthcare System , Little Rock, AR; Keith N. Humphreys, PhD MA, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (2):
- United States (2):
  - Central Arkansas Veterans Healthcare System , Little Rock, AR, Little Rock, Arkansas
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California

IPD SHARING:
Plan to Share IPD: Yes
Datasets meeting VA standards for disclosure to the public will be made available post-publication. Prior to distribution, a local privacy officer will certify that all datasets do not contain PHI. Final data sets will be maintained locally until enterprise-level resources become available for long-term storage and access. Guidance on request and distribution processes will be provided by ORD. Those requesting data will be asked to sign a Letter of Agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available following publication of the study results
Access Criteria: see above

REFERENCES:
- [Result] Cucciare MA, Marchant K, Benton C, Hildebrand D, Ghaus S, Han X, Thompson RG, Timko C. Connect To Care (C2C): protocol for two-site randomized controlled pilot trial to improve outcomes for patients with hazardous drinking and PTSD and/or depression symptoms. Addict Sci Clin Pract. 2023 Aug 17;18(1):50. doi: 10.1186/s13722-023-00403-z. PMID 37592359
- [Result] Cucciare MA, Benton C, Hildebrand D, Marchant K, Ghaus S, Han X, Williams JS, Thompson RG, Timko C. Adapting an Alcohol Care Linkage Intervention to US Military Veterans Presenting to Primary Care with Hazardous Drinking and PTSD and/or Depression Symptoms: A Qualitative Study. J Clin Psychol Med Settings. 2024 Jun;31(2):417-431. doi: 10.1007/s10880-023-09986-w. Epub 2023 Dec 15. PMID 38100057

DOCUMENTS (1):
  • Informed Consent Form (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT05023317/ICF_000.pdf